CLINICAL TRIAL: NCT05244304
Title: Phase 3, Multicenter, Randomized, Double-Masked, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Tinlarebant in the Treatment of Stargardt Disease in Adolescent Subjects
Brief Title: Phase 3, Randomized, Placebo-Controlled Study of Tinlarebant to Explore Safety and Efficacy in Adolescent Stargardt Disease
Acronym: DRAGON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Belite Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBS-008-CT03
Record Dates: First submitted 2022-01-20; First posted 2022-02-17 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Stargardt Disease 1
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Intervention Model Description: This is a Phase 3 randomized, double-masked, parallel group, multicenter study to evaluate the efficacy and safety of Tinlarebant 5 mg in the treatment of adolescent subjects with STGD1.
Who Masked: Participant, Investigator
Masking Description: Eligible subjects will be randomly assigned to begin treatment in 2:1 ratio to receive the study drug (either Tinlarebant 5 mg or matching placebo)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tinlarebant (Experimental): 5 mg tablet taken orally once a day
  Interventions: Drug: Tinlarebant
- Placebo (Placebo Comparator): Placebo tablets for tinlarebant 5 mg are prepared similarly but use microcrystalline cellulose, NF, in place of the active drug substance and will be identical in size and appearance.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tinlarebant — Tinlarebant drug substance is a white to off-white substance and is dispensed as a tablet for oral administration.
  Arms: Tinlarebant
Drug: Placebo — Not active drug
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to assesses the efficacy of tinlarebant in slowing the rate of growth of atrophic lesion(s) in adolescent subjects with STGD1

DETAILED DESCRIPTION:
Approximately 90 subjects will be enrolled in this study. Subjects will be assigned to study drug (tinlarebant 5 mg/placebo) with treatment period of upto 24 months with 28 days of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 12 to 20 years old, inclusive.
* Subject must have clinically diagnosed STGD1 (Stargardt disease 1) with at least 1 mutation identified in the ABCA4 gene.
* Subject must have a defined aggregate atrophic lesion size within 3 disc areas (7.62 mm2), as imaged by FAF in the study eye Subjects must have a BCVA of 20/200 or better for the study eye based on ETDRS letter score
* Subject and their parent(s) or legal guardian are willing to provide their consent on an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)/Human Research Ethics Committee (HREC)-approved informed consent form (ICF) prior to participating in any study-related procedures.
* Subject agrees to comply with all protocol requirements.

Exclusion Criteria:

* Any ocular disease other than Stargardt (STGD1) at baseline that, in the opinion of the investigator, would complicate assessment of a treatment effect.
* History of ocular surgery in the study eye in the last 3 months.
* Investigational drug use of any kind in the last 3 months or within 5 half-lives of the investigational drug, whichever is shorter.
* Any prior gene therapy.
* Vitamin A (retinol) deficiency as defined as a retinol serum level less than 20 mcg/dL (=0.7 μmol/L).

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
To measure change in atrophic lesion size (definitely decreased autofluorescence, DDAF) by fundus autofluorescence (FAF) photography from baseline | Baseline thru month 24

SECONDARY OUTCOMES:
To measure the change in retinal thickness assessed by spectral-domain optical coherence tomography (SD-OCT) from baseline | Baseline thru month 24
To measure the change in retinal morphology assessed by spectral-domain optical coherence tomography (SD-OCT) from baseline | Baseline thru month 24
To measure change in BCVA (Best Corrected Visual Acuity) score measured by the EDTRS method from baseline | Baseline thru month 24
To measure change in plasma concentration of RBP4 levels (μM) from baseline | Baseline thru month 24
The correlation between change in plasma RBP4 level and the rate of lesion size growth (definitely decreased autofluorescence, DDAF) by fundus autofluorescence (FAF) photography from baseline | Baseline thru month 24
To assess the systemic and ocular safety and tolerability of tinlarebant | Baseline thru month 24
  Frequency, duration, and severity of AEs

OTHER OUTCOMES:
To measure change in total decreased autofluorescence (DAF) by FAF photography from baseline | Baseline thru month 24
To measure change in questionably decreased autofluorescence (QDAF) by FAF photography from baseline | Baseline thru month 24
To measure change in quantitative autofluorescence (qAF) level from baseline | Baseline thru month 24
To measure change in retinal sensitivity by microperimetry from baseline | Baseline thru month 24

CONTACTS AND LOCATIONS:
Locations (19):
- United States (3):
  - Belite Study Site, Palo Alto, California
  - Belite Study Site, Minneapolis, Minnesota
  - Belite Study Site, Salt Lake City, Utah
- Australia (3):
  - Belite Study Site, Westmead, New South Wales
  - Belite Study Site, East Melbourne, Victoria
  - Belite Study Site, South Brisbane
- Belite Study Site, Ghent, Belgium
- China (2):
  - Belite Study Site, Beijing
  - Belite Study Site, Shanghai
- Belite Study Site, Paris, France
- Germany (2):
  - Belite Study Site, Bonn
  - Belite Study Site, Tübingen
- Belite Study Site, Kowloon, Hong Kong
- Belite Study Site, Nijmegen, Netherlands
- Belite Study Site, Basel, Switzerland
- Taiwan (2):
  - Belite Study Site, Taipei
  - Belite Study Site, Taoyuan
- United Kingdom (2):
  - Belite Study Site, London
  - Belite Study Site, Southampton

IPD SHARING:
Plan to Share IPD: No